CLINICAL TRIAL: NCT01181492
Title: Impact of CYP3A4*1G Polymorphism on Metabolism of Fentanyl in Chinese Patients Undergoing Lower Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: HuazhongU
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-08

CONDITIONS: Pain; Surgery
Keywords: gene polymorphism; CYP3A4; fentanyl; HPLC; Analgesics
MeSH Terms: conditions — Pain

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — 176 blood samples were extracted
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- *1/*1: Grouped by CYP3A4*1G polymorphism, wild-type homozygote
- *1/*1G: Grouped by CYP3A4*1G polymorphism,*1/*1G: mutant heterozygote
- *1G/*1G: Grouped by CYP3A4*1G polymorphism,*1G/*1G: mutant homozygote

SUMMARY:
Purpose: This study aimed to investigate the impact of CYP3A4*1G genetic polymorphism on metabolism of fentanyl in Chinese patients undergoing lower abdominal surgery. Methods: 176 patients receiving elective lower abdominal surgery under general anesthesia were recruited into this study. Genotyping of CYP3A4*1G was carried out by direct sequencing. The plasma fentanyl concentration was detected 30 min after anesthesia induction by high performance liquid chromatography-ultraviolet ray (HPLC-UV). The visual analog scale (VAS) was used for pain evaluation at rest during patient-controlled analgesia (PCA) treatment 0 h, 12 h and 24 h after operation. PCA fentanyl consumption and adverse effects were recorded during the first 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65 years
* Anesthesiologists (ASA) physical status I or II;
* With ±20% of ideal body weight;
* Received PCA administration;
* Agreed to participate the research

Exclusion Criteria:

* History of chronic pain;
* Psychiatric diseases;
* Diabetes mellitus;
* Severe cardiovascular diseases;
* Kidney or liver diseases;
* Alcohol or drug abuse (according to the criteria of DSM-IV);
* Pregnancy or at lactation period;
* Consumed drugs (1week) or foods (3 days) known to inhibit or induce the expression of CYP3A4 enzymes prior to surgery;
* Refused PCA administration;
* Disagree to participate to the research

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 176 Chinese patients receiving elective lower abdominal surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xianwei, MD, Study Director — Huazhong University of Science and Technology
Locations (1):
- 1. Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, from November 2008 to April 2010 a total of 176 patients were recruited in this study precedure.
Period: Overall Study
Arm/Group | *1/*1 | *1/*1G | *1G/*1G
Started | 103 | 66 | 7
Completed | 103 | 66 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | *1/*1 | *1/*1G | *1G/*1G | Total
Number analyzed (Participants) | 103 | 66 | 7 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 103 | 66 | 7 | 176
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.7) | 47.1 (10.1) | 42.3 (7.8) | 45.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 34 | 4 | 93
  Male | 48 | 32 | 3 | 83
Region of Enrollment [Number; unit: participants]
  China | 103 | 66 | 7 | 176

OUTCOME MEASURES:

1. Primary Outcome: CYP3A4*1G Polymorphism
Description: According to CYP3A4*1G polymorphism,patients are devided into three groups: *1/*1,*1/*1G,*1G/*1G
Time Frame: 48 hours after operation
Population: the number of participants for analysis was determined according to gene type of CYP3A4*1G polymorphism which was carried by participant.
Measure: Number; unit: participants
Arm/Group | *1/*1 | *1/*1G | *1G/*1G
Number analyzed (Participants) | 103 | 66 | 7
participants | 103 | 66 | 7

2. Secondary Outcome: The Visual Analog Scale 24 Hours Postoperative
Description: The visual analog scale (VAS) is used for pain evaluation at rest which from 0 to 10 (higher values represent morepain) during patient-controlled analgesia (PCA) treatment 24 h after operation
Time Frame: 24 hours after operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | *1/*1 | *1/*1G | *1G/*1G
Number analyzed (Participants) | 103 | 66 | 7
units on a scale | 3.7 (1.3) | 3.7 (1.1) | 3.4 (1.3)

3. Secondary Outcome: PCA Fentanyl Consumption
Description: PCA fentanyl consumption and adverse effects are recorded during the first 24 h after surgery.
Time Frame: 24 h after surgery
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | *1/*1 | *1/*1G | *1G/*1G
Number analyzed (Participants) | 103 | 66 | 7
μg | 395.0 (138.5) | 359.8 (120.2) | 247.1 (73.2)

ADVERSE EVENTS:
Arm/Group | *1/*1 | *1/*1G | *1G/*1G
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/66 | 0/7
Other Adverse Events (participants affected / at risk) | 0/103 | 0/66 | 0/7

LIMITATIONS AND CAVEATS:
The preoperative and postoperative data were not all integrallty recorded in a relative short period and entered into Excel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No